CLINICAL TRIAL: NCT01948921
Title: Meperidine as the Single Sedative Agent for Patients Expected to Have Poor Tolerance During Diagnostic Esophagogastroduodenoscopy.
Brief Title: Meperidine for Patients Expected to Have Poor Tolerance During Diagnostic Esophagogastroduodenoscopy.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dalin Tzu Chi General Hospital (Other)
Responsible Party: Principal Investigator, Yu-Hsi hsieh, Chief of Gastroenterology Endoscopy Suite, Dalin Tzu Chi General Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Diagnostic
Other Study IDs: DalinTCGH-hsieh-2013-3
Record Dates: First submitted 2013-09-19; First posted 2013-09-24 (Estimated); Last update posted 2017-03-20 (Actual); Status verified 2017-03

CONDITIONS: Patients Undergoing Diagnostic EGD
Keywords: EGD; tolerance; discomfort
MeSH Terms: interventions — Meperidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- placebo (Placebo Comparator): 1 ml normal saline will be given 5 minutes before EGD
  Interventions: Drug: placebo
- meperidine (Active Comparator): 25 mg intramuscular meperidine will be given 5 minutes before EGD
  Interventions: Drug: Meperidine

INTERVENTIONS:
Drug: placebo
  Arms: placebo
Drug: Meperidine
  Arms: meperidine

SUMMARY:
Our pilot results showed that meperidine reduce patient discomfort during EGD (esophagogastroduodenoscopy). But many patients can tolerate EGD well without any sedative agents. So the investigators target the use of meperidine on patients expected to have poor tolerance in this study, which includ young females with high anxiety level and patients with prior poor tolerance. The investigators test the hypothesis that meperidine improves tolerance and alleviates discomfort for patients expected to have poor tolerance during diagnostic EGD.

ELIGIBILITY:
Inclusion Criteria:

* female youger than 65 years with high anxiety level
* patients with previous poor tolerance of EGD

Exclusion Criteria:

* a therapeutic EGD
* sedation with other agents
* contraindication to Buscopan (hyoscine N-butylbromide) or meperidine
* American Society of Anesthesiology (ASA) risk Class 3 or higher, renal failure
* age less than 20 years or more than 80 years
* pregnancy
* refusal to provide written informed consent. All participants signed written informed consents

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2013-09; Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
discomfort score during esophageal intubation | 10 minutes
  self-reported discomfort score during esophageal intubation, assessed with a 0 to 10 (0 = none; 10 = unbearable) visual analog scale (VAS).

SECONDARY OUTCOMES:
patient discomfort score during the procedure | 10 minutes
patients satisfaction score | 10 minutes
patient tolerance score evaluated by the endoscopist | 10 minutes
endoscopist satisfaction score | 10 minutes

CONTACTS AND LOCATIONS:
Locations (1):
- Buddhist Dalin Tzu Chi General Hospital, Chiayi City, Taiwan, Taiwan

REFERENCES:
- [Background] Abraham NS, Fallone CA, Mayrand S, Huang J, Wieczorek P, Barkun AN. Sedation versus no sedation in the performance of diagnostic upper gastrointestinal endoscopy: a Canadian randomized controlled cost-outcome study. Am J Gastroenterol. 2004 Sep;99(9):1692-9. doi: 10.1111/j.1572-0241.2004.40157.x. PMID 15330904
- [Background] Hsieh YH, Lin HJ, Hsieh JJ, Tseng KC, Tseng CW, Hung TH, Leung FW. Meperidine as the single sedative agent during esophagogastroduodenoscopy, a double-blind, randomized, controlled study. J Gastroenterol Hepatol. 2013 Jul;28(7):1167-73. doi: 10.1111/jgh.12183. PMID 23431993
- [Background] Ishido S, Kinoshita Y, Kitajima N, Itoh T, Nishiyama K, Tojo M, Yano T, Inatome T, Fukuzaki H, Chiba T. Fentanyl for sedation during upper gastrointestinal endoscopy. Gastrointest Endosc. 1992 Nov-Dec;38(6):689-92. doi: 10.1016/s0016-5107(92)70565-3. PMID 1473671
- [Background] Laluna L, Allen ML, Dimarino AJ Jr. The comparison of midazolam and topical lidocaine spray versus the combination of midazolam, meperidine, and topical lidocaine spray to sedate patients for upper endoscopy. Gastrointest Endosc. 2001 Mar;53(3):289-93. doi: 10.1016/s0016-5107(01)70400-2. PMID 11231385